CLINICAL TRIAL: NCT03977402
Title: INST UNM 1521: Total Cancer Care Protocol: A Lifetime Partnership With Patients Who Have or May be at Risk of Having Cancer
Brief Title: Total Cancer Care Protocol: A Lifetime Partnership With Patients Who Have or May be at Risk of Having Cancer
Acronym: TCCP
Status: Recruiting | Type: Observational
Sponsor: New Mexico Cancer Research Alliance (Other)
Collaborators: H. Lee Moffitt Cancer Center and Research Institute (Other); Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: INST UNM 1521
Record Dates: First submitted 2019-05-08; First posted 2019-06-06 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Cancer; Cancer Risk
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Excess tissue, blood and/or fluids (normal and tumor; in the form of frozen and/or formalin fixed, paraffin-embedded tissue) removed from the patient following any extirpative surgical procedure (required as part of standard medical care) for future cancer research studies.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Biological specimen collection — Collection of blood, tissue, other biological samples and their associated data (survey data, medical records data, cancer registry data, and other related data) from patients with cancer or at risk of having cancer. This is not a treatment trial. It is a study designed to create a centralized data and tissue repository.
  Other Names: Medical chart review

SUMMARY:
The overall objective of this study is to ultimately develop an improved standard of cancer care by facilitating new cancer research, clinical trials, new technology, new informatics solutions, and "personalized medicine" for the University of New Mexico Comprehensive Cancer Center (UNMCCC) and the Oncology Research Information Exchange Network (ORIEN) Consortium of academic medical centers, community hospital systems, and other health care providers. To bring new translational research to the community, the ORIEN consortium has initiated the ORIEN Total Cancer Care Program (TCCP). The TCCP establishes a unique collection of blood, tissue, other biological samples and their associated data (survey data, medical records data, cancer registry data, and other related data) from thousands of patients with cancer or at risk of having cancer. This is not a treatment trial. It is a study designed to create a centralized data and tissue repository.

DETAILED DESCRIPTION:
Through this protocol, UNMCCC and its partners will establish and maintain a unique repository of blood, tissue, other biological samples and their associated data (survey data, medical records data, cancer registry data, and other related data) collected from thousands of patients 18 years of age or older who have cancer or are at risk of developing cancer. In this protocol, the investigators require the permission of patients to study their answers to survey questions that may be collected as part of their regular clinical care, permission to study their medical and related records, and permission to collect excess tissues removed at the time of planned surgery, an additional tumor sampling (needle passes) at the time of planned diagnostic biopsies, previously collected, stored tumor tissue (if available), blood, and/or other biological samples. Additional research tumor samples may be collected at the time of any diagnostic needle biopsy or endoscopic biopsy or, if available, patient tissue from a previous procedure will be obtained and utilized as needed. Clinical and related data will be collected on all patients from the time of initial entry into the study and will continue for life.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older.
* Has a diagnosis of cancer or is suspected of having cancer.
* Able to understand and sign the Informed Consent form directly.
* Pregnant women are permitted to be enrolled.

Exclusion Criteria:

* Prisoners

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients 18 years of age or older who have cancer or are at risk of developing cancer.
Sampling Method: Non-Probability Sample
Enrollment: 47500 (Estimated)
Dates: Start 2016-01-27 (Actual); Primary Completion 2036-12-31 (Estimated); Study Completion 2037-12-31 (Estimated)

PRIMARY OUTCOMES:
Amount of clinical patient demographic data collected for a repository linked to clinical data for long-term research use. | up to 20 years
  Establish a longitudinal clinical data repository that will contain information about patient demographics collected via surveys and questionnaires.
Amount of clinical patient medical treatment and outcome data collected via medical histories for long-term research use | up to 20 years
  Establish a longitudinal clinical data repository that will contain information about medical treatments and patient outcomes collected via medical chart review and patient medical histories.
Number of biospecimens collected for a tissue repository linked to clinical data for long-term research use | up to 20 years
  Establish a longitudinal tissue repository that will contain tissues (blood, tumor tissue) and other biological samples and associated clinical data collected from consenting patients.

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Andritsos, MD, Principal Investigator — University of New Mexico Cancer Center
Locations (1):
- University of New Mexico Comprehensive Cancer Center, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: Yes
As an ORIEN member institution, UNMCCC will share limited data with the ORIEN consortium, including patient identifiers, collected from patients with known or suspected cancer. UNMCCC may also distribute any blood, tissue samples, or other biological samples with protected health information according to the Information Warehouse (IW) TCCP honest broker policy and UNM Human Tissue Repository (HTR).
Time Frame: Unknown at this time
Access Criteria: ORIEN consortium membership